CLINICAL TRIAL: NCT04713228
Title: Prospective Case-Control Study of Cardiovascular Changes in Pregnancy Related Hypertensive Disorders
Acronym: ARTSEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Indu Poornima, Director, Section of Cardiovascular Prevention, AHN; Professor of Medicine, Drexel University College of Medicine, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-128
Record Dates: First submitted 2021-01-06; First posted 2021-01-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Pregnant with Pre-eclampsia (Experimental): There will be an initial 'Pregnancy' visit within 7-10 days of the screening visit, when the subject will undergo an echocardiogram, have the vascular compliance measurements and will have blood drawn for measurement of serum biomarkers. The second study visit will be the '6-8 weeks post-partum' visit when the echocardiogram and vascular compliance will be re-measured, along with assessment of vitals and medication history. The third study visit will be 6-7 months post partum where there is a collection of a clinical questionnaire, demographics, vitals, chart review, echocardiogram and vascular compliance will be re-measured.
  Interventions: Device: ARTSENS Pen
- Pregnant with gestational hypertension (Experimental): There will be an initial 'Pregnancy' visit within 7-10 days of the screening visit, when the subject will undergo an echocardiogram, have the vascular compliance measurements and will have blood drawn for measurement of serum biomarkers. The second study visit will be the '6-8 weeks post-partum' visit when the echocardiogram and vascular compliance will be re-measured, along with assessment of vitals and medication history. The third study visit will be 6-7 months post partum where there is a collection of a clinical questionnaire, demographics, vitals, chart review, echocardiogram and vascular compliance will be re-measured.
  Interventions: Device: ARTSENS Pen
- Pregnant without Hypertension - Control (Active Comparator): There will be an initial 'Pregnancy' visit within 7-10 days of the screening visit, when the subject will undergo an echocardiogram, have the vascular compliance measurements and will have blood drawn for measurement of serum biomarkers. The second study visit will be the '6-8 weeks post-partum' visit when the echocardiogram and vascular compliance will be re-measured, along with assessment of vitals and medication history. The third study visit is not applicable to the control group.
  Interventions: Device: ARTSENS Pen

INTERVENTIONS:
Device: ARTSENS Pen — ARTerial Stiffness Evaluation for Noninvasive Screening

SUMMARY:
This is a research study to understand the changes in the heart and the cardiovascular system that may occur in women who develop high blood pressure during pregnancy.

DETAILED DESCRIPTION:
Upon Enrollment in this study, participants will go through two scans along with some blood test and other assessments. The first scan is a sonogram of the heart called an echocardiogram, and another scan is done using the investigational ARTSENS device that will be used to measure stiffness of the walls in the arterial blood vessel for indications of inflammation damage. ARTSENS device is not approved for use in the United States. It is expected that we will enroll 50 people in this study. The entire study is expected to last 2 years. Participation will be for approximately 9 months.

ELIGIBILITY:
Case Inclusion Criteria:

1. Adult females age > 18 years
2. Must be able to read and understand English and consent for themselves
3. Must have a singleton pregnancy and a diagnosis of preeclampsia or gestational hypertension
4. Must be willing and able to come to West Penn Hospital for post-partum visits at 6-8 weeks and then at 6-7 months.

Case Exclusion Criteria:

1. Prior history of hypertension
2. Multiple pregnancies
3. Other comorbidities such as congenital heart disease, dialysis dependent renal failure, heroin abuse, cocaine abuse, pulmonary hypertension, congestive heart failure, autoimmune conditions such as SLE or severe lung disease.
4. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Control Inclusion Criteria:

1. Adult females age > 18 years
2. Must be able to read and understand English and consent for themselves
3. Must have a singleton pregnancy and not have a prior or current diagnosis of hypertension
4. Must be willing and able to come to West Penn Hospital for post-partum visits at 6-8 weeks.

Control Exclusion Criteria:

1. Prior history and/or current diagnosis of hypertension
2. Multiple pregnancies
3. Other comorbidities such as congenital heart disease, dialysis dependent renal failure, heroin abuse, cocaine abuse, pulmonary hypertension, congestive heart failure, autoimmune conditions such as SLE or severe lung disease.
4. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrolling pregnant women
Enrollment: 12 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Function measured as Left ventricular ejection fraction (LVEF) | 6 months
  Measurement: LVEF is expressed as a % and Global longitudinal strain measurement also expressed as %.
  Measurements tools: two dimensional echocardiography and strain imaging with speckle tracking echocardiography
Change in Diastolic function | 6 months
  Measurement: E/E' velocity; This is a ratio and there is no unit for measurement.
  Measurement tools: Pulse Doppler echocardiography
Change in vascular compliance | 6 months
  Measurement:
  Pulse strain elasticity (Ep) expressed as kPa, Arterial stiffness Beta which is an index without units.
  Measurement tool: Arterial waveforms captured with the ARTSENS device
Change in vascular stiffness | 6 months
  Measurement: Beta which is an index without units
  Measurement tool: Arterial waveforms captured with the ARTSENS device

SECONDARY OUTCOMES:
Correlation of left ventricular ejection fraction (LVEF) with troponin and proBNP | 3 months
  Cardiac measurements: LVEF is in %, Troponin is ng/ml, proBNP is pmol/L
  Measurement tool:
  LVEF is measured with 2D echocardiography, proBNP and Troponin is measured by blood sample assessing biomarker alterations that could predict cardiovascular damage.
Correlation of vascular compliance and stiffness | 3 months
  Measurement: Pulse strain elasticity (Ep) expressed as kPa, Arterial stiffness Beta which is an index without units, E/E' is a ratio
  Measurement tool: Arterial waveforms captured with the ARTSENS device and Doppler Echo.

CONTACTS AND LOCATIONS:
Overall Officials: Indu Poornima, MD, Principal Investigator — Allegheny Health Network Research Insititute
Locations (1):
- West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published; patient identifiers will not be used in the research publications.